CLINICAL TRIAL: NCT05605652
Title: Evaluation of Leveling and Alignment of Maxillary Anterior Teeth Assisted With Micro-osteoperforations:A Comparative Clinical Study.
Brief Title: Evaluation of Leveling and Alignment of Maxillary Anterior Teeth Assisted With MOPs :A Comparative Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Omar Mohamed abd elsalam abo donia, Omar Abodonia, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 660/301
Record Dates: First submitted 2022-10-31; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Crowding of Anterior Maxillary Teeth
MeSH Terms: interventions — morpholinopropane sulfonic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): leveling and alignment will be commenced without micro- osteoperforations
- Experimental group (Experimental): Flapless micro-osteoperforations will be performed interproximally on the alveolar bone equidistant between upper right canine to upper left canine at every interdental alveolar bone except at the midline
  alveolar bone to prevent trauma to the soft tissue frenum before placing the initial leveling archwire.
  Interventions: Procedure: microosteoperforations

INTERVENTIONS:
Procedure: microosteoperforations — Flapless micro-osteoperforations will be performed interproximally on the alveolar bone equidistant between upper right canine to upper left canine at every interdental alveolar bone except at the midline
  alveolar bone to prevent trauma to the soft tissue frenum before placing the initial leveling archwire.
  Other Names: MOPs
  Arms: Experimental group

SUMMARY:
The aim of the study will be directed to evaluate the effect of micro-osteoperforation on orthodontic tooth movement during leveling and alignment of the maxillary anterior teeth.

DETAILED DESCRIPTION:
The current study will be conducted on a group of orthodontic patients attending the out patients clinic, Orthodontic Department, Faculty of Dental Medicine (Boys), AL- Azhar University, Cairo

The patient will be randomly assigned into two equal groups:

1. Experimental group: Flapless micro-osteoperforations will be performed interproximally on the alveolar bone equidistant between upper right canine to upper left canine at every interdental alveolar bone except at the midline

   alveolar bone to prevent trauma to the soft tissue frenum before placing the initial leveling archwire.
2. Control group: leveling and alignment will be commenced without micro- osteoperforations.

ELIGIBILITY:
Inclusion Criteria:

* 1. Class 1 skeletal pattern with normal facial proportions. 2. Patients with age range between 13 -19 years. 3. Moderate crowding of maxillary anterior region assessed by Little Irregularity Index (LII) that require treatment with fixed appliance using non extraction approach.

  4. All permanent teeth erupted (excluding 3rd molars). 5. No previous orthodontic treatment. 6. Good oral hygiene with no previous periodontal surgery.

Exclusion Criteria:

* 1. Transverse and/or vertical skeletal dysplasia or craniofacial malformation. 2. Retained primary or missing permanent teeth in the maxillary anterior area. 3. Poor oral hygiene 4. Present or history of periodontal diseases. 5. Physical or mental disability. 6. Systemic diseases or regular use of medications that could interfere with orthodontic tooth movement.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
• Alignment progress was evaluated on 3D digital model taken before inserting the 1st archwire and then at all subsequent visits using (LII). | 2months-6months
  • Alignment progress was evaluated on 3D digital model taken before inserting the 1st archwire and then at all subsequent visits using (LII).
• Overall time needed to complete leveling and alignment of maxillary anterior segment | 2months -6months
  • Overall time needed to complete leveling and alignment of maxillary anterior segment was calculated by the number of days between day of inserting the 1st archwire and at the end of the leveling and alignment stage.
• Alignment improvement percentage | 2months -6months
  • Alignment improvement percentage was calculated by dividing the amount of change in the LII value at a specific time point (calculated by subtracting the LII value at T1, T2, or T3 from the LII value at T0) by LII value at T0.

CONTACTS AND LOCATIONS:
Overall Officials: Raafat GH Mohamad, Asst Prof, Study Chair — Department of orthodontics, Faculty of Dental Medicine (Boys-Cairo), Al-Azhar University; Ahmed A El-Awady, Lecturer, Study Director — Department of orthodontics, Faculty of Dental Medicine (Boys-Cairo), Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Nasr City, Egypt